CLINICAL TRIAL: NCT07042477
Title: An Integrated, Virtual and On-Demand Solution to Avoid ED Utilization
Brief Title: Integrated Telemedicine Program Evaluation
Acronym: ITP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Amir Goren, Principal Investigator, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-0554
Record Dates: First submitted 2025-06-18; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Behavioral Intervention; Emergency Department Visits; Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Telemedicine Program (Experimental): Patients will be invited to participate in the integrated telemedicine program through text, email, and/or phone calls.
  Interventions: Behavioral: Integrated Telemedicine Program
- Control (No Intervention): Patients will receive only standard care and will receive no invitation to participate in the integrated telemedicine program.

INTERVENTIONS:
Behavioral: Integrated Telemedicine Program — The integrated telemedicine program is short-term bridge support provided by a virtually accessible team, including a behavioral health provider (Health Psychologist or Licensed Clinical Social Worker [LCSW]) and Community Health Worker (CHW). Once stabilized, members transition from bridge support to ongoing care with a Geisinger Health System Primary Care Provider and Behavioral Health Provider.
  Arms: Integrated Telemedicine Program

SUMMARY:
This project will evaluate a virtual, on-demand telemedicine program for High emergency department (ED) utilizers with comorbid physical health conditions and behavioral health correlates. Researchers will randomize patients to have either full access to the full intervention (treatment group) or to receive only standard care (control group). Analyses will be intent-to-treat. The primary outcome is the number of ED visits 120 days after the first Best Practice Alert (BPA) firing.

The research team plans to enroll 3200 patients in this study. However, randomization may end due to system constraints on December 31, 2025 before reaching that target. This sample provides 80% power to detect a 35% relative reduction in ED utilization using a two-tailed test with an alpha of .15, assuming 40% compliance with the program.

ELIGIBILITY:
Patient presents to the ED and meets the following criteria:

Inclusion Criteria:

* 18+ years old
* 4+ Geisinger ED visits in the last 6 months
* Geisinger Health Plan (GHP) insurance member
* Has a Geisinger PCP
* Patient is being seen at one of the following facilities: Geisinger Lewistown Hospital, Geisinger Medical Center, Geisinger Bloomsburg Hospital, Geisinger Jersey Shore Hospital, Geisinger Community Medical Hospital, Geisinger Wyoming Valley, Geisinger Medical Center Muncy, Geisinger Shamokin Ach Hospital, Geisinger South Wilkes Barre

Exclusion Criteria:

* Patient being seen in departments determined ineligible by the study team
* Patient is diagnosed with alcohol and substance-related disorders
* Patient is going to receive inpatient care
* Patient is coded in the ED as Level 1 (i.e., seeking life-saving measures)
* Patient has an Intellectual Disability or Traumatic Brain Injury
* Patient is actively seeing a BH provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3200 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Emergency Department Visits | within 120 days of the initial BPA firing
  Number of emergency department visits

OTHER OUTCOMES:
Health-related quality of life (HRQoL) | Within 120 days of randomization
  HRQoL will be measured via the RAND Short Form 36 (36-item questionnaire) administered each BH visit. A high score indicates a better health state or functioning. The lowest and highest possible scores are 0 and 100 respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Geisinger Clinic, Danville, Pennsylvania, United States